CLINICAL TRIAL: NCT04903080
Title: Phase 1 Trial of Autologous HER2-specific CAR T Cells in Pediatric Patients With Refractory or Recurrent Ependymoma
Brief Title: HER2-specific Chimeric Antigen Receptor (CAR) T Cells for Children With Ependymoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: Texas Children's Cancer Center (Other); Baylor College of Medicine (Other); National Cancer Institute (NCI) (NIH); American Lebanese Syrian Associated Charities (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-059; UM1CA081457 (NIH); NCI-2021-06710 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-059 (Other: Pediatric Brain Tumor Consortium); PBTC-059 (Other: CTEP)
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Ependymoma
MeSH Terms: conditions — Ependymoma

STUDY DESIGN:
Intervention Model Description: This study includes two groups: a safety cohort and a surgical cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (HER2 CAR T cells), Phase I Arm (Experimental): Patients receive lymphodepletion chemotherapy with cyclophosphamide IV daily on Days -7 to -6 and fludarabine IV daily on Days -5 to -1. Patients receive HER2 CAR T cells IV on Day 0. Treatment repeats every 8 to 12 weeks for 2 additional cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: HER2 Specific CAR T Cell
- Treatment (HER2 CAR T cells), Surgical Arm (Experimental): Patients receive lymphodepletion chemotherapy with cyclophosphamide IV daily on Days -7 to -6 and fludarabine IV daily on Days -5 to -1. Patients receive HER2 CAR T cells IV on Day 0 followed by surgical tumor resection 4-6 weeks following HER2 CAR T cell infusion. Treatment repeats every 8 to 15 weeks for 2 additional cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: HER2 Specific CAR T Cell

INTERVENTIONS:
Biological: HER2 Specific CAR T Cell — HER2 CAR (Chimeric Antigen Receptor) T cells are T cells that have been genetically engineered to target the protein HER2 for the treatment of cancer.

SUMMARY:
This is a Phase I study to evaluate the safety profile of a type of immune therapy called HER2 CAR T cells (short for HER2 chimeric antigen receptor T cells). In addition to looking for side effects, we will study how well this treatment works against a brain tumor called ependymoma that has come back after treatment (recurrent) or has not responded well to treatment (progressive) in children. The HER2 CAR T cells used in this trial are made from the patient's own blood. A new gene, called the HER2 CAR, will be inserted into patient's T cells to allow them recognize a protein on the tumor called HER2. These HER2-specific CAR T cells may be able to target and kill ependymoma tumors that express HER2. This research is also studying how doable it is to provide this type of CAR T cell treatment to children being treated at different hospitals.

DETAILED DESCRIPTION:
PBTC-059 is a multicenter, Phase I and Surgical study of the treatment HER2-specific CAR T cells for patients with refractory or recurrent ependymoma.

Phase I

The primary objectives of the Phase I study are to determine the safety of intravenous injection of HER2-specific CAR T cells after lymphodepleting chemotherapy, and to evaluate the multicenter feasibility of administering up to three infusions of HER2-CAR T cells after lymphodepletion.

Patients will receive one infusion of HER2psecific CAR T cells after lymphodepleting chemotherapy. Following recovery from their first treatment (no earlier than 8 weeks and no later than 12 weeks), patients will resume treatment with HER2-specific CAR T cells for up to 2 infusions after lymphodepleting chemotherapy if they meet laboratory parameters.

The length of time on study for patients enrolled on the Phase I study is anticipated to be 9 months on treatment. Patients will then be followed for 15 years after treatment.

Surgical Study

The objective of the Surgical study is to evaluate the post-treatment tumor tissue for presence of HER2-specific CAR T cells administered intravenously in children undergoing surgical resection. The surgical study will be initiated following completion of the safety evaluation period of 6 patients treated in the Phase I study.

Once the surgical study is open for enrollment, all patients who have clinical indication for surgery, except those needing urgent surgery, will be eligible for enrollment to the surgical study. Patients will receive one infusion of HER2-specific CAR T cells after lymphodepleting chemotherapy 4-6 weeks before surgical resection of their tumor, at which time samples will be taken for analysis. Following recovery from surgery (no earlier than 8 weeks and no later than 15 weeks), patients will resume treatment with HER2-specific CAR T cells for up to 2 infusions if they meet laboratory parameters.

The first patient in the surgical study will complete a 6-week safety evaluation period prior to enrollment of the subsequent patient. The length of time on study for patients enrolled on the Surgical study is anticipated to be 10 months on treatment. Patients will then be followed for 15 years after treatment.

Dosing

All patients on Phase I and Surgical study will receive HER2 CAR T cells at a patient-specific dose level 1 (8x10^7 CAR-positive T cells/m^2) for infusion. The cell dose will be based on the patient weight and height obtained by the treating institution at the time of procurement. For patients whose BMI is greater than 95th percentile for given age and sex, the Body surface area (BSA) will be calculated using the ideal body weight.

In the event that dose level 1 is found to have excessive toxicity, three additional doses of CAR T cells at dose level -1 (5x10^7 CAR-positive T cells/m^2) will be made to be used in the event that dose de-escalation occurs before a patient is enrolled for treatment.

ELIGIBILITY:
Criteria for Screening

1. Tumor

   Patient must have a diagnosis of ependymoma that is recurrent or progressive. All tumors must have histologic verification either at the time of diagnosis or recurrence.
2. Prior Therapy

   Patient must have received standard of care therapy including maximal safe surgical resection followed by local adjuvant radiation therapy prior to enrollment.
3. Adequate Pre-trial Tumor Tissue

   Patient must have adequate pre-trial tumor material available to determine HER2 status. Tumor tissue from the most recent resection or biopsy of recurrent disease in preferred. If unavailable, tumor tissue from prior recurrences or from the time of initial diagnosis is acceptable.

   a. One exception will be patients who have previously received HER2-directed therapy (including but not limited to trastuzumab); these patients will need evaluation of tumor HER2 status after stopping treatment due to the possibility of HER2 downregulation or loss.

   Tumor biopsy will not be performed for the purpose of HER2 screening. Patients will not be eligible for screening on PBTC-059 if tumor tissue is not available or inadequate for HER2 testing. Tumor screening by Immunohistochemistry (IHC) will be done centrally using the testing method validated at Texas Children's Hospital. Sample for screening must be shipped within 7 days of enrollment for screening.
4. Known HIV Positivity

   Patients that are known to be HIV-positive are ineligible due to the unknown safety and efficacy of infusing these patients with CAR T cells genetically modified using retroviral vectors. Additionally, the immunosuppression used for treatment in this study will pose an unacceptable risk.
5. Age

   Patient must be ≥ 1 but ≤ 21 years of age at the time of screening consent.
6. Screening Consent

   The patient or parent/guardian can understand the consent and is willing to sign a written informed consent document according to institutional guidelines. Age- and developmentally appropriate assent should be obtained as required by institutional guidelines.
7. Potential Eligibility for Study Treatment Enrollment

Patients are screened for this trial should be reasonably anticipated to meet the criteria for treatment described in Section 3.3 if their tumor is HER2-positive.

Criteria for Procurement

All subjects must meet following inclusion and exclusion eligibility criteria at the time of peripheral blood procurement for manufacturing the HER2 CAR T-cell product. No exceptions will be given. All clinical and laboratory evaluations to establish eligibility for procurement must be done within 14 days prior to enrollment. See Section 6.1 for details of laboratory requirements and planning of procurement blood collection date.

Procurement Inclusion Criteria

1. Tumor

   Patient must have been screened and determined to have a diagnosis of a HER2-positive recurrent or progressive ependymoma.
2. Performance Score

   Karnofsky Performance Scale (KPS for > 16 years of age) or Lansky Performance Score (LPS for ≤ 16 years of age) (Appendix C) assessed within one week of procurement must be ≥ 60%. Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score provided the neurological deficit is stable as described in Section 3.3.1.7.
3. Prior Therapy

   Patients must have received last dose of cytotoxic chemotherapy greater than 21 days preceding the date of enrollment for procurement.
4. Organ Function

   Patient must have adequate organ and bone marrow function as defined below:
   1. Peripheral absolute neutrophil count (ANC) > 1.0 x 109 cells/L
   2. Platelet count ≥ 75 100 x 109 cells/L (unsupported, defined as no platelet transfusion within 4 days)
   3. Hemoglobin ≥ 8 g/dL (may receive red blood cell transfusions)
   4. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) for age
   5. Alanine transaminase (ALT /SGPT) and Aspartate aminotransferase(AST/SGOT) ≤ 3 x institutional upper limit of normal (ULN) for age
   6. Serum creatinine < 1.5 x institutional upper limit of normal for age and gender. Patients that do not meet the criteria but have a 24-hour Creatinine Clearance or Glomerular filtration rate (GFR) (radioisotope or iothalamate) ≥ 70 mL/min/1.73 m2 are eligible.
   7. Pulmonary Function

      * Oxygen saturation as measured by pulse oximetry is ≥ 93% on room air.
5. Concomitant Medication

   Patients who are receiving systemic corticosteroids must be on a stable or decreasing dose for at least two weeks prior to procurement, and corticosteroid dose must be less than or equal to dexamethasone 0.75 mg/m2/day (or equivalent). Use of topical, ocular, intranasal, or inhaled corticosteroids are permitted.
6. Procurement Consent

   The patient or parent/guardian can understand the consent and is willing to sign a written informed consent document according to institutional guidelines. Age- and developmentally appropriate assent should be obtained as required by institutional guidelines.
7. Potential Eligibility for Study Enrollment

Patients whose blood samples have been successfully procured for this trial should be reasonably anticipated to meet the criteria for treatment described in Section 3.3 and to begin treatment within 180 days from the date of procurement. The treatment slot will not be held beyond the specified 180 days, and such patients may not be able to receive treatment on this study depending on slot availability.

Procurement Exclusion Criteria

1. Known HIV Positivity

Patients who are known to be HIV-positive are ineligible due to the unknown safety and efficacy of infusing these patients with CAR T cells genetically modified using retroviral vectors. Additionally, the immunosuppression used for treatment in this study will pose an unacceptable risk.

Criteria for Treatment

All Phase I (Stratum 1) and Surgical (Stratum 2) subjects must meet following inclusion and exclusion eligibility criteria at the time of enrollment for treatment. No exceptions will be given. Imaging studies must be done within 14 days prior to enrollment. All other clinical and laboratory evaluations to establish eligibility for treatment must be done 7 days prior to enrollment.

Treatment Inclusion Criteria

1. Diagnosis

   Patients with a histologically confirmed diagnosis of HER2 positive ependymoma that is recurrent or progressive. Histologic verification may be from time of diagnosis or time of recurrence. In cases where there is question of recurrence, histologic verification, or verification of progression on follow up imaging is required prior to enrolling for protocol treatment.
2. Disease Status

   Phase I (Stratum 1) - Patients must have evaluable disease to be eligible. Evaluable disease includes either measurable OR non-measurable disease, defined as follows:
   1. Measurable disease (enhancing or non-enhancing tumor):

      * at least 1 cm, or
      * at least two times (in both perpendicular diameters) the MRI slice thickness, plus the interslice gap.
   2. Non-measurable disease (tumor that is too small to be accurately measured):

      * less than 1 cm in at least one perpendicular dimension, or
      * less than two times the MRI slice thickness, plus the interslice gap.

   Note: Leptomeningeal disease is considered non-measurable but evaluable.

   Surgical Study (Stratum 2) - Patients with measurable disease (Section 3.3.1.2.1) in whom tumor resection is clinically indicated and feasible after the CAR T cell infusion.
3. Age

   Patient must be ≥ 1 but ≤ 22 years of age at the time of enrollment for treatment.
4. HER2 CAR T cell product

   The patient must have, at a minimum, one prescribed dose of the cryopreserved, autologous HER2 CAR T cell product available for infusion.
5. Prior Anti-neoplastic Therapy

   Cytotoxic chemotherapy: Patients must not have received cytotoxic chemotherapy for at least 28 days prior to study enrollment for treatment and must have recovered from the acute treatment related toxicities (defined as < grade 1 if not defined in eligibility criteria; excludes alopecia) prior to entering this study.

   Biological, targeted, or investigational agents (anti-neoplastic): Patients must have a period of at least 28 days from the last receipt of said drug and must have recovered from all acute toxic effects.
   1. For agents that have known acute adverse events occurring beyond 28 days after administration, this period must be extended beyond the time during which adverse events are known to occur.

   Monoclonal antibodies, checkpoint inhibitors, and other agents with known prolonged half-lives: Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent ≥ 28 days prior to study enrollment.

   Adoptive cellular therapies: Patient must have recovered from any acute toxicity potentially related to the cellular product and received their last dose of the cellular product at least 90 days prior to study enrollment. (Note: Patients who have previously received an adoptive cellular therapy may continue long-term follow up evaluations per the prior study's evaluation schedule as needed for assessment of long-term toxicities including genotoxicity.)

   Radiation: Patients must have had their last fraction of:

   a. Craniospinal irradiation, whole brain radiation, total body irradiation or radiation to >50% of pelvis or spine ≥ 3 months prior to enrollment (90 days) prior to enrollment.

   b. Focal palliative irradiation to the tumor ≥ 42 days prior to enrollment. c. Patients who receive tumor-directed radiation (non-palliative) should have confirmed disease progression on the imaging study done at least 6 weeks after the completion of the last fraction of radiation.

   Surgery: Patients must have not had surgery within 14 days of enrollment for treatment and must have adequate wound healing and recovered from other acute effects from surgery. One exception is the placement of central venous catheter which will be allowed at any time point until treatment initiation on the study.
6. Growth Factors

   Patients must be off all colony-forming growth factor(s) for at least 7 days prior to enrollment (e.g., filgrastim, sargramostim, or erythropoietin). 14 days must have elapsed if the patient received a long-acting formulation.
7. Corticosteroids

   Patients who are receiving systemic corticosteroids must be on a stable or decreasing dose for at least 14 days prior to enrollment for treatment, and corticosteroid dose must be less than or equal to dexamethasone 0.5 mg/m2/day (or equivalent) during the 14 days preceding enrollment. Use of topical, ocular, intranasal, or inhaled corticosteroids are permitted.
8. Neurologic Status

   In patients with neurological deficits, deficits should be stable for a minimum of 7 days prior to enrollment. A baseline detailed neurological exam should clearly document the neurological status of the patient at the time of enrollment for treatment on the study.

   Patients with seizure disorders may be enrolled if seizures are well controlled.
9. Performance Status

   Karnofsky Performance Scale (KPS for > 16 years of age) or Lansky Performance Score (LPS for ≤ 16 years of age) (Appendix C) assessed within one week of enrollment must be ≥ 60%. Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
10. Organ Function

    Patients must have adequate organ and bone marrow function as defined in Section 3.2.1.4.
11. Pregnancy Prevention

    Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study.
12. Informed Consent

The patient or parent/guardian can understand the consent and is willing to sign a written informed consent document according to institutional guidelines. Age- and developmentally appropriate assent should be obtained as required by institutional guidelines.

1. Patients who meet eligibility criteria per Section 3.3.1.2.1 must be enrolled using Phase I treatment consent (Stratum 1).
2. Patients who meet eligibility criteria per Section 3.3.1.2.2 must be enrolled using Surgical Study treatment consent (Stratum 2).

Treatment Exclusion Criteria

1. Patients with Bulky Tumors on Imaging Studies

   Bulky tumors will be defined as those:
   1. > 6 cm in single maximum dimension, or
   2. tumor causing uncal herniation or mass effect leading to midline shift with or without symptoms or signs of impending herniation or
   3. obstruction to Cerebrospinal fluid (CSF) flow.
2. Infratentorial tumors with symptoms or signs arising from brain stem involvement by the tumor. Patients with stable cranial nerve deficit(s) secondary to prior surgery will not be excluded.
3. Surgical Study (Stratum 2): Patients who have urgent need for surgical resection of tumor.
4. Pregnancy or Breast-feeding

Pregnant women or nursing mothers are excluded from this study.

a. Female patients of childbearing potential must have a negative serum or urine pregnancy test within 7 days of start of enrollment for treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Pregnant or breast-feeding women are excluded from this study because there is an unknown but potential risk of adverse events to the fetus or the nursing infant with the use of T cells genetically modified to express HER2 CAR. Pre-clinical studies in mice demonstrate the target antigen HER2 is necessary for normal fetal development of cardiac trabeculae, cranial sensory ganglia, and motor neuron development.75 Additionally, the lymphodepleting chemotherapy drugs fludarabine and cyclophosphamide are both Pregnancy Class D drugs.

4. Concurrent Illness

Patients with active autoimmune disease, documented history of autoimmune disease/syndrome, or any other condition that requires ongoing systemic steroids or systemic immunosuppressive agents, except a. Patients with vitiligo or resolved asthma/atopy b. Patients with hypothyroidism stable on hormone replacement or Sjogren's syndrome c. Patients requiring physiologic doses of corticosteroids (up to 0.5 mg/m2/day dexamethasone equivalent)

History of or ongoing pneumonitis or significant interstitial lung disease

Ongoing or active uncontrolled infection

Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the opinion of the investigator, would compromise the patient's ability to tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results.

Patients with any of the following cardiac diseases

1. New York Heart Association (NYHA) functional class III or IV
2. Clinically significant cardiac arrhythmia including, but not limited to, Torsade de pointes or requiring a pacemaker
3. Left ventricular ejection fraction below 50% as determined by echocardiography (ECHO)

Known HIV positivity

a. HIV-positive patients are ineligible due to the unknown safety and efficacy of infusing these patients with CAR T cells genetically modified using retroviral vectors. Additionally, the immunosuppression used for treatment in this study will pose an unacceptable risk.

5. Concomitant Medications

Patients who are receiving any other anti-cancer or investigational drug therapy are ineligible.

Patients who have received the last vaccination of a live vaccine ≤ 30 days prior to enrollment are ineligible.

1. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and must meet timeline for live vaccine.

Herbal preparations/medications (except for vitamins) including, but not limited to: St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, black cohosh, and ginseng. Patients should stop using all herbal medications and dietary supplements at least 7 days prior to enrollment.

6. Inability to participate

Patients who in the opinion of the investigator are unwilling or unable to return for required follow-up visits or obtain follow-up studies required to assess toxicity to therapy or to adhere to drug administration plan, other study procedures, and study restrictions.

7. Allergy

Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition (murine protein-containing products, Dimethylsulfoxide (DMSO), or dextran 40).

Ages: 1 Year to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2043-07-20 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with Dose-Limiting Toxicity (DLT) in Phase I Arm | Up to 42 days following the first CAR T cell infusion
  DLT is defined as an adverse event that is at least possibly attributed to the investigational agent (HER2 CAR T cells) that occurs during the dose-finding period (the first 42 days following the first CAR T cell infusion) regardless of expectedness with a few exceptions, for which Section 6.4 of the protocol provides more details. All patients in Safety/Feasibility cohort who received at least 1 dose of HER2 CAR T cells are included in the assessment.
Number of Subjects with Dose-Limiting Toxicity (DLT) in Surgical Arm | Up to 42 days following the first CAR T cell infusion
  DLT is defined as an adverse event that is at least possibly attributed to the investigational agent (HER2 CAR T cells) that occurs during the dose-finding period (the first 42 days following the first CAR T cell infusion) regardless of expectedness with a few exceptions, for which Section 6.4 of the protocol provides more details. All patients in Surgical cohort who received at least 1 dose of HER2 CAR T cells are included in the assessment.
Percentage of Subjects whose Treatment Delivery Meets Feasibility Criteria | Approximately 3 months after enrollment for treatment
  Assessment of feasibility is in the context of conducting an investigator-initiated (not industry sponsored) multi-institutional trial of CAR T cells. This would specifically include the feasibility of manufacturing the cells at one center and shipping them to other sites for administration and the infusion process. If more than 25% of patients cannot be treated as intended due to manufacturing, shipping or administration related causes (jointly considered as feasibility criteria), this would be considered unacceptable. If the treatment is not delivered as intended due to one or more manufacturing, shipping, or administration related causes, this instance will be counted as feasibility failure for that subject.

SECONDARY OUTCOMES:
Expansion and Persistence of HER2 CAR T Cells at First Infusion in patients who received this treatment | Approximately 3 months after enrollment for treatment
  Frequency of HER2-specific CAR T cells is measured at first infusion in treated subjects. Data are summarized at pre- and post-infusion time points to evaluate their expansion and persistence.
Expansion and Persistence of HER2 CAR T Cells at Second Infusion in patients who received this treatment | Approximately 7 months after enrollment of treatment
  Frequency of HER2-specific CAR T cells is measured at second infusion in treated subjects. Data are summarized at pre- and post-infusion time points to evaluate their expansion and persistence.
Expansion and Persistence of HER2 CAR T Cells at Third Infusion in patients who received this treatment | Approximately 10 months after enrollment for treatment
  Frequency of HER2-specific CAR T cells is measured at third infusion in treated subjects. Data are summarized at pre- and post-infusion time points to evaluate their expansion and persistence.
Presence of intra-tumoral HER2 CAR T Cells following First Infusion in Surgical Arm | Approximately 3 months after enrollment for treatment
  Frequency of HER2-specific CAR T cells is measured at first infusion in subjects in Surgical cohort. Data are summarized at pre- and post-infusion time points to evaluate their expansion and persistence.
Presence of HER2 CAR T Cells following Second Infusion in Surgical Arm | Approximately 6 months after enrollment for treatment
  Frequency of HER2-specific CAR T cells is measured at second infusion in subjects in Surgical cohort. Data are summarized at pre- and post-infusion time points to evaluate their expansion and persistence.
Presence of HER2 CAR T Cells following Third Infusion in Surgical Arm | Approximately 9 months after enrollment for treatment
  Frequency of HER2-specific CAR T cells is measured at third infusion in subjects in Surgical cohort. Data are summarized at pre- and post-infusion time points to evaluate their expansion and persistence.
Best antitumor Response of Infused HER2 CAR T Cells in Phase I Arm | Up to 15 years from the initiation of protocol treatment
  Proportion of subjects with complete response (CR) or partial response (PR) is calculated. Patients in Safety/Feasibility cohort who received at least 1 dose of CAR T cells are considered. CR refers to complete resolution of all evaluable tumor and mass effect maintained for at least 4 weeks. PR refers to for measurable disease a greater than or equal to 50% reduction in tumor size by bi-dimensional measurement maintained for at least 4 weeks.
Best Antitumor Response of Infused HER2 CAR T Cells in Surgical Arm | Up to 15 years from the initiation of protocol treatment
  Proportion of subjects with complete response (CR) or partial response (PR) or clinical complete response (CCR) is calculated. Patients in Surgical cohort who received at least 1 dose of CAR T cells are considered. CR refers to complete resolution of all evaluable tumor and mass effect maintained for at least 4 weeks. PR refers to for measurable disease a greater than or equal to 50% reduction in tumor size by bi-dimensional measurement maintained for at least 4 weeks. CR and PR are for subjects with measurable disease. CCR is for subjects who do not have measurable disease.
Event-free Survival (EFS) | Up to 2 years from the initiation of protocol treatment
  2-year EFS is estimated for all eligible subjects who initiated the conditioning regimen. EFS is defined as the time interval between date of initiation of protocol treatment and minimum date of documentation of disease progression, second malignancy, death due to any cause, or date of last follow-up.
Overall Survival (OS) | 2 years from the initiation of protocol treatment
  2-year OS is estimated for all eligible subjects who initiated the conditioning regimen. OS is defined as the time interval between date of initiation of protocol treatment and date of death due to any cause or date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Meenakshi Hegde, MD, Study Chair — Baylor College of Medicine
Locations (13):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Pittsburgh Children's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Texas Children's Cancer Center, Houston, Texas
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No